CLINICAL TRIAL: NCT00958412
Title: A Randomized, Double-blind Study Evaluating the Safety and Efficacy of Proellex® in the Treatment of Premenopausal Women With Symptomatic Endometriosis-extension Study
Brief Title: Study Evaluating the Safety and Efficacy of Proellex® in the Treatment of Endometriosis-extension Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Repros stopped the study for safety and FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPE-201 EXT
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pelvic pain; Oral progesterone blocker
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proellex® (Experimental): 25 mg Proellex®
  Interventions: Drug: Proellex®

INTERVENTIONS:
Drug: Proellex® — one (1) 25 mg capsule daily
  Other Names: CDB-4124

SUMMARY:
ZPE-201 Extension of treatment

DETAILED DESCRIPTION:
This is an extension of the phase II, three-arm, parallel design, dose-ranging, placebo-controlled, randomized, double-blind, multicenter study in which placebo or one (1) of two (2) dose levels of Proellex® was administered once-daily for four (4) months.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects treated in the ZPE-201 study will be allowed to enter the extension study.
* Subjects who withdrew from ZPE-201 due to lack of treatment efficacy will also be invited to participate.

Exclusion Criteria:

* All other subjects

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02-28 (Actual); Primary Completion 2009-08-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (8):
- United States (8):
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - Compass Clinical Research, San Ramon, California
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Physicians for Women, Cary, North Carolina
  - HWC Women's Research Center, Miamisburg, Ohio
  - Clinical Trials of Texas/Institute for Women's Health, San Antonio, Texas
  - Clinical Trials of Texas/Seven Oaks Women's Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Proellex: Proellex: one (1) 25 mg capsule daily Study was terminated prematurely and no data is available
Period: Overall Study
Arm/Group | Proellex
Started | 18
Completed | 0
Not Completed | 18
Not completed — Study prematurely terminated | 18

BASELINE CHARACTERISTICS:
Population: A total of 18 participants were randomized; study prematurely terminated.
Arm/Group | Proellex®
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Incidence of Adverse Events (AEs) and Safety of Proellex® Administered Once Daily
Description: Number of participants who experienced 1 or more adverse event.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Proellex®
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Proellex®: Proellex®: one (1) 25 mg capsule daily No data available
Arm/Group | Proellex®
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Proellex® (N=18)
Seasonal Allergies (Immune system disorders) | 1
1.5 % decrease femur bone density (Investigations) | 1
abnormal labs (Investigations) | 1
cervical tenderness (Reproductive system and breast disorders) | 1
Crying (Nervous system disorders) | 1
Cystic Left Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decrease in Bone mineral Density (Investigations) | 2
Decreased bone Mineral Density in the Lumbar Spine (Investigations) | 2
Decreased Libido (Reproductive system and breast disorders) | 1
Elevated ALT (Investigations) | 1 — ALT (Alanine Transaminase)
Elevated AST (Investigations) | 1 — AST (Aspartate Transaminase)
exacerbation migraine (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hot Flashes (Vascular disorders) | 4
Influenza (Infections and infestations) | 1
Irregular Heart Beat (Cardiac disorders) | 1
joint pain (Musculoskeletal and connective tissue disorders) | 1
Left Cystic Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Left hip bone mineral density decreased (Investigations) | 1
left lower quadrant pain (Gastrointestinal disorders) | 1
left ovarian complex cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lumbar Spine Bone Mineral Density Decreased (Investigations) | 1
Mood Swings (Nervous system disorders) | 2
Right lower quadrant abdomen pain (Gastrointestinal disorders) | 1
Right ovarian complex cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
right ovarian cyst 1.5cm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Right Paraovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
sinus infection (Infections and infestations) | 1
skin rash (Skin and subcutaneous tissue disorders) | 1
vaginal discharge (Reproductive system and breast disorders) | 1
verruca vulgaris (Infections and infestations) | 1
weight gain (Investigations) | 1
Yeast Infection (Infections and infestations) | 1
sexual desire loss (Reproductive system and breast disorders) | 1
insomnia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights